CLINICAL TRIAL: NCT04806009
Title: Evaluating an Online Mindfulness-Based Intervention for Individuals With Insomnia in China: A Randomized Controlled Trial
Brief Title: Evaluating an Online Mindfulness-Based Intervention for Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Chen Pan, Principal Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CentralSouthU2021
Record Dates: First submitted 2021-03-07; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Insomnia, Primary
Keywords: insomnia; mindfulness-based intervention; Cognitive Behavioral Therapy for insomnia; online
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Mindful Living With Insomnia (MLWI)' Intervention via WeChat mini-program (Experimental): Participants in the Intervention Group will receive the MLWI Intervention after follow the WeChat mini-program. The MLWI Intervention was developed and presented by the Principle Investigator (PI) who is a psychiatrist and have completed the Training of Mindfulness Facilitation (TMF) program at the Mindful Awareness Research Center of University of California, Los Angeles.
  Interventions: Behavioral: 'Mindful Living With Insomnia (MLWI)' Intervention via WeChat mini-program
- 'Cognitive Behavioral Therapy for insomnia (CBT-I)'via WeChat mini-program (Active Comparator): Participants in the Control Group will receive CBT-I after follow the WeChat mini-program. The CBT-I was developed and presented by a researcher who is a psychiatrist/psychologist and have many years' experiences in CBT.
  Interventions: Behavioral: 'Cognitive Behavioral Therapy for insomnia (CBT-I)'via WeChat mini-program

INTERVENTIONS:
Behavioral: 'Mindful Living With Insomnia (MLWI)' Intervention via WeChat mini-program — The MLWI Intervention involves 12 sessions over 6 weeks course, 2 sessions a week and 0.5 hours per session. Two new sessions of online lessons will be updated weekly in the 6 weeks. Each session is consisted of theoretical lecture, mindfulness practices, sharing common difficulties and coping way during mindfulness practices and homework assignment in the form of video or audio. The Mindfulness practices embedded in the intervention include mindful breathing, mindful body scan, mindful dealing with thoughts and emotions, mindful meditation, mindful movement, and daily life mindfulness. In the intervention, the participants will also receive sleep hygiene education.Participants in the Intervention Group will receive the MLWI Intervention after follow the WeChat mini-program.
  Arms: 'Mindful Living With Insomnia (MLWI)' Intervention via WeChat mini-program
Behavioral: 'Cognitive Behavioral Therapy for insomnia (CBT-I)'via WeChat mini-program — The CBT-I involves 12 sessions over 6 weeks course, 2 sessions a week and 0.5 hours per session. Two new sessions of online lessons will be updated weekly in the 6 weeks. Each session is consisted of theoretical lecture, cognitive or behavioral regulation techniques, sharing common difficulties and coping way during mindfulness practices and homework assignment in the form of video or audio.Participants in the Control Group will receive CBT-I after follow the WeChat mini-program.
  Arms: 'Cognitive Behavioral Therapy for insomnia (CBT-I)'via WeChat mini-program

SUMMARY:
Insomnia has significantly negative impact on work, quality of life, psycho-somatic health on individuals and imposes substantial economic burdens on society. Mindfulness-based interventions (MBIs) have shown its efficacy in the treatment of insomnia, however the effect of online MBIs need more studies to verify. This study aims to compare the effectiveness of an online MBI named 'Mindful Living With Insomnia (MLWI)' to online CBI-I for insomnia.

DETAILED DESCRIPTION:
This will be an online based, randomized, controlled trial. Investigators will recruit 1000 participants, and will randomize and allocate participants 1:1 to the 'Mindful Living With Insomnia (MLWI)' group (n=500) and the 'CBT-I' group (n=500). The Intervention will involve 12 sessions over 6 weeks course, 2 sessions a week and 0.5 hours per session. The primary outcome will be sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI), severity of insomnia symptoms assessed by the Insomnia Severity Index (ISI), and sleep parameters recorded using Mi Smart Band. The secondary outcomes include perceived stress, anxiety, depression, and mindfulness. Outcomes will be evaluated at baseline, the end of the intervention period, and at a 3-month follow-up. Analysis of covariance, regression analysis, χ2 test, t-test, Pearson's correlations will be applied in data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 59 years old
2. Being able to read and write Chinese
3. PSQI exceeding 5 at screening
4. Being able to access online services
5. Willing to participate in the study

Exclusion Criteria:

1. Unable to communicate
2. With somatic disorders
3. With mental disorders except for insomnia disorder
4. Being treated with pharmacotherapy
5. Significant current mindfulness practices (>15 minutes/ day)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
change of sleep quality | Outcomes will be evaluated at baseline, the end of the 6-week Intervention Period, and at a 3-month follow-up
  The 19-item Pittsburgh Sleep Quality Index (PSQI) measured sleep quality subjectively and assesses sleep disturbances during the past month on a 4-point Likert scale of 0 -3.A lower global PSQI score indicates better sleep quality.

SECONDARY OUTCOMES:
change of perceived stress | Outcomes will be evaluated at baseline, the end of the 6-week Intervention Period, and at a 3-month follow-up
  Perceived stress will be assessed by Perceived Stress Scale (PSS). The PSS has 14 items. Items are rated on a 5-point Likert-type scale, with higher total scores indicating higher perceived stress (0-13, low perceived stress; 14-26, moderate perceived stress; 27-40, high perceived stress).
change of depression | Outcomes will be evaluated at baseline, the end of the 6-week Intervention Period, and at a 3-month follow-up
  Depression will be assessed using the Patient Health Questionnaire (PHQ-9). The PHQ-9 consists of 9 items and all items are rated on a 4-point scale (0 = never; 3 = always), with higher total scores indicating more severe depression. Cutoffs are 5, 10, 15, and 20 for mild, moderate, moderately severe, and severe depression, respectively. The standard cut-off score of 10 or greater maximized combined sensitivity and specificity.
change of mindfulness | Outcomes will be evaluated at baseline, the end of the 6-week Intervention Period, and at a 3-month follow-up
  Mindfulness level will be assessed using Five Facets Mindfulness Questionnaire (FFMQ).FFMQ consists of 39 items which range from 1 (never or very rarely true) to 5 (very often or always true). The higher the total score, the more mindful the individual is.
change of anxiety | Outcomes will be evaluated at baseline, the end of the 6-week Intervention Period, and at a 3-month follow-up
  Anxiety will be assessed using the Generalized Anxiety Disorder Questionnaire (GAD-7). The GAD-7 has 7 items for assessing the level of general anxiety.All items are rated on a 4-point scale (0 = never; 3 = always), with higher total scores indicating higher levels of anxiety, and a cutoff score >6 is recommended to identify anxiety symptoms.
change of severity of insomnia symptoms | Outcomes will be evaluated at baseline, the end of the 6-week Intervention Period, and at a 3-month follow-up
  The 7-item ISI assesses the current severity of insomnia symptoms, sleep dissatisfaction, daytime impacts, and distress concerning difficulties with sleep on a 5-point Likert scale (0 = never; 4 = always). Total scores range from 0 to 28. Cutoffs are 8, 15, 22 for subthreshold, moderate and severe insomnia respectively.
change of sleep duration and quality | Outcomes will be evaluated at baseline, the end of the 6-week Intervention Period, and at a 3-month follow-up
  Digital biomarker data such as sleep duration and quality, and daytime activity will be assessed by Mi Wristband.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Pan, Dr, Principal Investigator — The Third Xiangya Hospital,Central South University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan C, Tie B, Yuwen W, Su X, Deng Y, Ma X, Wu Y, Liao Y, Kong L, Zhang Y, Li Z, Pan Q, Tang Q. 'Mindfulness Living with Insomnia': an mHealth intervention for individuals with insomnia in China: a study protocol of a randomised controlled trial. BMJ Open. 2022 Feb 15;12(2):e053501. doi: 10.1136/bmjopen-2021-053501. PMID 35168972